CLINICAL TRIAL: NCT04297046
Title: Ultrasound-guided Transversus Abdominis Plane Block and Quadratus Lumborum Block as Preventive Analgesia in Total Abdominal Hysterectomy With Pfannenstiel Incision: a Prospective, Randomized Trial
Brief Title: Ultrasound-guided Two Different Type Blocks for Pain Relief in Totalabdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Canan Yılmaz, principal investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-7/9
Record Dates: First submitted 2020-02-28; First posted 2020-03-05 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Ultrasonography
Keywords: Nerve block; analgesia; pain management
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: After general anesthesia was given to the participant, the blocks were made. The participant did not know the type of block made to him.The outcomes assessor evaluating the participants after the surgery does not know the type of block made to the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB for total abdominal hysterectomy (Active Comparator): Quadratus lumborum block (QLB) was performed bilaterally with 0,3 ml/kg 0.25% bupivacaine (maximum dose 3 ml/kg) solution injection on each side.Combine patient-controlled intravenous analgesia(same as PCA for TAH arm).
  Interventions: Device: PCA (patient controlled analgesia)
- TAPB for total abdominal hysterect0my (Active Comparator): The transversus abdominis plane block (TAPB)was performed bilaterally with 0.3 ml/kg of 0.25% bupivacaine (maximum dose 3 ml/kg) solution . Combine patient-controlled intravenous analgesia(same as PCA for TAH arm).
  Interventions: Device: PCA (patient controlled analgesia)

INTERVENTIONS:
Device: PCA (patient controlled analgesia) — Intravenous Patient-Controlled Analgesia was used for postoperative pain control with a bolus dose of 25 mg Tramadol and a lockout interval of 20 min. The pain was evaluated at different times after the operation, both at rest and movement (Dynamic VAS) at the 0., 2., 6., 12. hours and 24h later. All patients received 1 g iv paracetamol 8 hourly intervals regularly. 75 mg im diclofenac sodium was given as rescue analgesic.

SUMMARY:
Effective analgesia after total abdominal hysterectomy is important for faster recovery and preventing complications which depend to pain. A multimodal and preventive approach is preferred to ensure adequate analgesia and to avoid side effects due to high doses of analgesics. The hypothesis was that the Quadratus Lumborum block (application of local anesthetics to the side of the abdomen) would be superior to Transversus Abdominis Plane block (application of local anesthetics in front of the abdomen) for analgesia before abdominal incision in total abdominal hysterectomy. The primary goal of the study was to evaluate the feasibility of ultrasound-guided Transversus Abdominis Plane block and Quadratus Lumborum block. The secondary goal was to evaluate postoperative adverse effects and patient satisfaction.

DETAILED DESCRIPTION:
The study protocol was approved by the Local Ethics Committee. Written informed consent was obtained from each patient. The study was carried out in accordance with The Code of Ethics of the Declaration of Helsinki. The study was conducted between April 2017 - July 2017 with a prospective, randomized, double-blind design on 62 patients who had undergone total abdominal hysterectomy with Pfannenstiel incision. American Society of Anesthesiologist (ASA) II-III, patients between the ages of 18-75 were included in the study. The participants with bleeding diathesis, those who could not communicate (mental disorder, language problem, etc.), those with allergies to the drugs used, those who did not wish to participate in the study, and those who had an infection in the block area were excluded from the study. The participants were divided into 2 groups with the sealed envelope technique preoperatively Transversus Abdominis Plane Block Procedure Before the surgical procedure, the muscles were screened at the umbilicus plain/mid-axillary line with the ultrasound using a linear probe while the participants in the supine position. The skin, subcutaneous adipose tissue, external oblique muscle, internal oblique muscle, transversus abdominis muscle, and peritoneum were visualized. The block needle was advanced in the posterolateral direction with the in-plain approach. 0.3 ml/kg of 0.25% bupivacaine was administered bilaterally into the space between the internal oblique muscle and the transversus abdominis muscle.

Transmuscular Quadratus Lumborum Block Procedure Quadratus lumborum muscle could be recognized with ultrasound via the convex probe was transversally attached above iliac crest at the midaxillary line while the patients were in the lateral decubitus position. The point of injection with a block needle in transmuscular Quadratus Lumborum Block is between the anterior border of Quadratus lumborum muscle and psoas major muscles. A transmuscular Quadratus Lumborum Block was performed bilaterally with 0,3 ml/kg 0.25% bupivacaine solution injection on each side.

ELIGIBILITY:
Inclusion Criteria:

* Undergone total abdominal hysterectomy with Pfannenstiel incision
* American Society of Anesthesiologist (ASA) I-III
* Patients between the ages of 18-65

Exclusion Criteria:

* Patients with bleeding diathesis
* Patients who could not communicate (mental disorder, language problem, etc.)
* Patients with allergies to the drugs used
* Patients who did not wish to participate in the study
* Patients who had an infection in the block area

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
iv PCA tramadol consumption | 24 hours
  tramadol consumption up to 24 hours
intraoperatively fentanyl use | during operation
  Total intraoperative fentanyl dose
The Visual analogue Scale (VAS) | 24 hours
  The Visual Analogue Scale was used to measure the severity of postoperative pain (0= No pain, 10= The worst possible pain) up to 24 hours. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
postoperative adverse effects | 24 hours
  nausea,vomiting, hypertension and hypotension incidences
patient and surgeon satisfaction: scores | 24 hours
  The patient and surgeon satisfaction score (0= Not satisfied, 4= Very satisfied) were recorded. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Yilmaz, Principal Investigator — Medical Doctor of Anesthesiology Department
Locations (1):
- Bursa Yuksek Ihtisas Education and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No